CLINICAL TRIAL: NCT04150250
Title: A Phase 2a Randomized, Single-Center, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Preliminary Efficacy of Oral iOWH032 Against Cholera Diarrhea in a Controlled Human Infection Model
Brief Title: Cholera Anti-Secretory Treatment Trial
Acronym: CAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: University of Maryland, Baltimore (Other); Pharmaron (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRG-032-PO-2-01-USA
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-02

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera | interventions — IOWH-032; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iOWH032 (Experimental): On Day 1, participants were challenged with 10^6 colony-forming units (CFU) of freshly-harvested wild-type V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever occurred first, participants received oral iOWH032 500 mg tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
  Interventions: Drug: iOWH032; Other: V. cholerae Challenge; Drug: Antibiotics
- Placebo (Placebo Comparator): On Day 1, participants were challenged with 10^6 CFU of freshly-harvested wild-type V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever occurred first, participants received oral matching iOWH032 placebo tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
  Interventions: Drug: Placebo; Other: V. cholerae Challenge; Drug: Antibiotics

INTERVENTIONS:
Drug: iOWH032 — Anti-secretory synthetically manufactured small molecule designed to inhibit the cystic fibrosis transmembrane conductance regulator chloride channel.
  Arms: iOWH032
Drug: Placebo — Oral tablets matching iOWH032 on taste, appearance, dissolution time with the same excipients but no active ingredients.
  Arms: Placebo
Other: V. cholerae Challenge — Freshly-harvested, wild-type Vibrio (V.) cholerae El Tor Inaba strain N16961,10^6 cfu suspended in 30 mL of sodium bicarbonate solution ingested orally.
Drug: Antibiotics — Antibiotic therapy may include:
  * Ciprofloxacin 500 mg, twice daily;
  * Azithromycin 500 mg, once daily (for those persons who are allergic to fluoroquinolones);
  * Doxycycline 300 mg, once daily (for those persons who are allergic to fluoroquinolones)

SUMMARY:
This trial was designed to assess safety and preliminary efficacy of oral doses of iOWH032 on diarrhea output and clinical symptoms after a cholera challenge in healthy adult participants.

DETAILED DESCRIPTION:
The study consists of a screening phase, an inpatient containment period with challenge with Vibrio cholerae on Day 1 followed by treatment with iOWH032 or placebo and a post-challenge observation period until discharge, an outpatient follow-up period of at least 28 days, and a final follow-up (by telephone) 6 months post-challenge (Day 180) for the collection of serious adverse events.

Participants will be randomized 1:1 to receive either iOWH032 500 mg every 8 hours for three days or matching placebo. Blinded therapeutic dosing will start at the onset of diarrhea or by 48 hours after ingesting the challenge inoculum of V. cholerae. The observation and management of cholera diarrhea and symptomatology will occur on an inpatient isolation research ward over a duration of approximately 11 days, including a three-day course of antibiotics to treat all participants prior to discharge from the inpatient unit.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and provide written informed consent
2. Healthy male and female adults, age 18 to 44 years (inclusive), without clinically significant medical history, physical or clinical laboratory abnormalities (as per protocol-defined acceptable ranges), and protocol-defined abnormal electrocardiogram results at screening
3. All women must have a negative serum pregnancy test at screening and one day prior to challenge.
4. Agreement by participants to use an adequate method of contraception* during the study and for 4 weeks before and after the challenge.
5. Able to pass a written examination (comprehension assessment test) with a score of ≥ 70%, in order to demonstrate their comprehension of this study. If a participant scores at least 50%, then they will be given one more opportunity to re-test after further re-education.
6. Willing and able to comply with the study requirements and procedures.

   * Adequate contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label; includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 4 weeks prior to study enrollment), or women who have intercourse limited to men who underwent vasectomy.

Exclusion Criteria:

1. Clinically significant history of immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease, anal or rectal disorders, neurologic disease,
2. Current nicotine use or drug, alcohol abuse within the past 6 months
3. Recipient of bone marrow or solid organ transplant
4. Use of systemic chemotherapy in the past 5 years
5. Has a malignancy (excluding localized non-melanoma skin cancers) or lymphoproliferative disorders diagnosed or treated within the past 5 years
6. Received or plans to receive systemic immunosuppressive therapy, radiation therapy, parenteral or high-dosage inhaled steroids (> 800 µg/day of beclomethasone dipropionate or equivalent) within 6 months prior to the enrollment through 28 days after challenge
7. Have a history of hospitalization for psychiatric illness, suicide attempt, or confinement for danger to self or others, within the past 10 years. Participants with a psychiatric disorder (not meeting exclusion criteria, e.g., attention-deficit hyperactivity disorder) that is controlled for a minimum of 3 months and the investigator has determined that the participant's mental status will not compromise the participant's ability to comply with protocol requirements may be enrolled
8. Have an elevated blood pressure, systolic ≥ 150 mmHg or diastolic ≥ 90 mmHg, before challenge
9. Taking any of the the protocol-defined drugs that are metabolized by CYP2C9 or any of the following psychiatric medications: aripiprazole, carbamazepine, chlorpromazine, chlorprothixene, clozapine, divalproex sodium, fluphenazine, haloperidol, lithium carbonate, lithium citrate, loxapine, mesoridazine, molindone, olanzapine, perphenazine, pimozide, quetiapine, risperidone, thioridazine, thiothixene, trifluoperazine, triflupromazine, or ziprasidone
10. History of Guillain-Barré Syndrome
11. Too low or too high a body mass index (BMI < 18.5 or > 39)
12. Has an abnormal stool pattern defined as fewer than 3 stools per week or more than 2 stools per day within the past 6 months, and any loose stools (grade 3 or higher) during the 1-2 day acclimation period before challenge
13. Has regularly used laxatives in the past 6 months
14. Has a history of eating disorders (e.g. anorexia or bulimia) within the past 10 years
15. Known allergy or previous severe adverse effect to all of the following antibiotics: ciprofloxacin (or quinolones), azithromycin and doxycycline.
16. Previously received a licensed or investigational cholera vaccine, within 10 years
17. History of cholera or enterotoxigenic Escherichia coli (ETEC) infection (lab-confirmed natural infection or experimental challenge), within 10 years
18. Travel to a cholera-endemic area in the past 5 years
19. Pregnant or nursing
20. Positive serology for human immunodeficiency virus (HIV), hepatitis B antigen, or hepatitis C antibody
21. Protocol-defined clinically abnormal 12-lead electrocardiogram (ECG) at screening in the judgment of the Investigator, or based on the formal 12-lead ECG reading by a cardiologist; history of any cardiac abnormalities, including conduction abnormalities such as Wolff-Parkinson-White, dysrhythmias, or coronary artery disease
22. Presence of a clinically significant abnormality on physical examination, including (but not limited to): pathologic heart murmur, lymphadenopathy, hepatosplenomegaly, large abdominal scar of unclear origin
23. Has poor venous access, defined as the inability to obtain screening blood tests after three attempts
24. Currently on, or plans to be on, antibiotics (e.g., doxycycline) within 14 days prior to challenge and through 28 days after challenge
25. Presence of an acute illness or fever (> 100.4°F) within 72 hours of admission to the inpatient Clinical Research Unit
26. Taking any prescription or over-the-counter medications that contain aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), antacids, proton pump inhibitors (PPIs), anti-diarrheals, etc. within 72 hours prior to challenge
27. Received an investigational product within 30 days prior to randomization (90 days prior to randomization for monoclonal antibodies) or planned to participate in another research study involving an investigational product during the conduct of this study
28. Participants must not have donated blood in 8 weeks prior to study entry and agreed to not donate blood during and for 4 weeks following their active participation in this study
29. Lack of ability to fully understand the informed consent
30. Any other condition(s) that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erdem R, Ambler G, Al-Ibrahim M, Fraczek K, Dong SD, Gast C, Mercer LD, Raine M, Tennant SM, Chen WH, de Hostos EL, Choy RKM. A Phase 2a randomized, single-center, double-blind, placebo-controlled study to evaluate the safety and preliminary efficacy of oral iOWH032 against cholera diarrhea in a controlled human infection model. PLoS Negl Trop Dis. 2021 Nov 18;15(11):e0009969. doi: 10.1371/journal.pntd.0009969. eCollection 2021 Nov. PMID 34793441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 healthy adults were enrolled at one clinical research site in the United States. Participants were confined in an inpatient isolation research ward for a duration of approximately 11 days until discharge criteria were met.
Pre-assignment Details: Participants were randomized in a 1:1 ratio stratified by blood type status (O vs. Non-O) to receive either iOWH032 500 mg every 8 hours for three days or matching placebo.
Groups:
- iOWH032: On Day 1, participants were challenged with 10^6 colony-forming units (CFU) of freshly-harvested wild-type V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever was first, participants received oral iOWH032 500 mg tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
- Placebo: On Day 1, participants were challenged with 10^6 CFU of freshly-harvested wild-type V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever was first, participants received oral matching iOWH032 placebo tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
Period: Overall Study
Arm/Group | iOWH032 | Placebo
Started | 23 | 24
Completed | 23 | 22
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- iOWH032: On Day 1, participants were challenged with 10^6 CFU of freshly-harvested wild-type V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever was first, participants received oral iOWH032 500 mg tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
- Total: Total of all reporting groups
Arm/Group | iOWH032 | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (6.15) | 32.3 (5.97) | 32.1 (6.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 5 | 7
  Black or African American | 21 | 19 | 40
Blood Type [Count of Participants; unit: Participants]
  Type O | 12 | 13 | 25
  Non-O | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Diarrheal Stool Output Rate
Description: Diarrheal stool output rate is defined as the total volume of diarrheal stools (in mL, Grade 3 and above) divided by the number of hours between initiation of study drug (iOWH032 or placebo) and initiation of antibiotic therapy.
  Stools were graded based on consistency as follows:
  * Grade 1 - well formed (normal stool, does not take the shape of the container)
  * Grade 2 - soft (normal stool, does not take the shape of the container)
  * Grade 3 - thick liquid (diarrhea, takes the shape of the container readily)
  * Grade 4 - opaque watery diarrhea
  * Grade 5 - rice water diarrhea (clear watery)
  The definition of diarrhea is a grade 3 or higher stool.
Time Frame: Day 1 - Day 5 (up to first dose of antibiotic therapy)
Population: Randomized participants who received at least one dose of study drug (iOWH032 or placebo) and with indication of cholera infection (diarrheal stool output of Grade 3 or higher) within 48 hours of challenge.
Measure: Median (Inter-Quartile Range); unit: mL/hour
Groups:
- iOWH032: On Day 1, participants were challenged with 10^6 CFU V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever occurred first, participants received oral iOWH032 500 mg tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
- Placebo: On Day 1, participants were challenged with 10^6 CFU V. cholerae. At the onset of diarrhea, or at 48 hours after challenge, whichever occurred first, participants received oral matching iOWH032 placebo tablets every 8 hours for 3 days. Participants received a 3-day course of antibiotics starting 4 days post-challenge, or sooner if the participant met the criterion for severe cholera diarrhea.
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
mL/hour | 25.42 [7.2 to 65.9] | 32.57 [14.7 to 53.0]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.2254, Van Elteren test — The threshold to define success on the primary efficacy endpoint at the final analysis is one-sided alpha = 0.0238; Stratified by blood type group (O vs. Non-O); Difference in Median = -7.1, 95% CI 2-sided [-30.9 to 28.6]

2. Primary Outcome: Diarrheal Stool Output Rate Including Participants With Symptom Onset After 48 Hours
Description: Stools were graded based on consistency as follows:
  * Grade 1 - well formed (normal stool, does not take the shape of the container)
  * Grade 2 - soft (normal stool, does not take the shape of the container)
  * Grade 3 - thick liquid (diarrhea, takes the shape of the container readily)
  * Grade 4 - opaque watery diarrhea
  * Grade 5 - rice water diarrhea (clear watery)
  The definition of diarrhea is a grade 3 or higher stool. For participants with symptom onset within 48 hours of challenge diarrheal stool output rate is defined as the total volume of diarrheal stools (mL, Grade 3 and above) divided by the number of hours between initiation of study product dosing and initiation of antibiotic therapy.
  For participants with symptom onset after 48 hours diarrheal stool output rate is defined as the total volume of diarrheal stools (mL, Grade 3 and above) divided by the number of hours between onset of symptoms and initiation of antibiotic therapy.
Time Frame: Day 1 - Day 5 (up to first dose of antibiotic therapy)
Population: Randomized participants who received at least one dose of study drug (iOWH032 or placebo) and with indication of cholera infection (diarrheal stool output of Grade 3 or higher) after challenge.
Measure: Median (Inter-Quartile Range); unit: mL/hour
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 20 | 23
mL/hour | 25.42 [6.3 to 63.8] | 29.22 [12.5 to 49.6]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.2751, Van Elteren test; Stratified by blood type group; Difference in Median = -3.8, 95% CI 2-sided [-26.3 to 27.4]

3. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events
Description: A serious adverse event (SAE) is any adverse event that resulted in any of the following outcomes:
  1. Death
  2. A life-threatening event.
  3. Required inpatient hospitalization or prolongation of existing hospitalization
  4. Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  5. Congenital abnormality or birth defect
  6. Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant and/or requires medical or surgical intervention to prevent one of the outcomes listed in the above definition of serious adverse event.
Time Frame: Day 1 - Day 180
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 23 | 24
Participants | 0 | 1

4. Secondary Outcome: Percentage of Participants With Moderate to Severe Diarrhea With Onset Within 48 Hours Following Cholera Challenge
Description: The percentage of participants with moderate to severe diarrhea with onset within 48 hours following cholera challenge.
  Diarrhea was defined as a grade 3 or higher stool based on the following scale:
  * Grade 1 - well formed (normal stool, does not take the shape of the container)
  * Grade 2 - soft (normal stool, does not take the shape of the container)
  * Grade 3 - thick liquid (diarrhea, takes the shape of the container readily)
  * Grade 4 - opaque watery diarrhea
  * Grade 5 - rice water diarrhea (clear watery)
  Diarrheal stools (Grade 3-5) were graded for severity according to the following: Mild: ≤ 3 liters loose stools; Moderate: > 3 liters loose stools; Severe: > 5 liters loose stools.
Time Frame: Day 1 - Day 5 (up to first dose of antibiotic therapy)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
percentage of participants | 43.8 [19.8 to 70.1] | 55.0 [31.5 to 76.9]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.5145, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, stratified by blood type group; Difference = -11.3, 95% CI 2-sided [-44.1 to 21.6]

5. Secondary Outcome: Attack Rate of Any Diarrhea Following Cholera Challenge
Description: Attack rate of any diarrhea following cholera challenge is defined as the number of participants with 2 or more loose stools (Grade 3-5) totaling > 200 mL or 1 loose (Grade 3-5) stool > 300 mL, respectively, with onset within 48 hours of cholera challenge.
Time Frame: Day 1 - Day 5 (up to first dose of antibiotic therapy)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
percentage of participants | 93.8 [69.8 to 99.8] | 100.0 [83.2 to 100.0]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.2636, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, stratified by blood type group; Difference = -6.3, 95% CI 2-sided [-18.1 to 5.6]

6. Secondary Outcome: Area Under the Curve (AUC) of Diarrheal Stool Volume Between Challenge Dose and Initiation of Antibiotics
Description: The AUC of diarrheal stool volume and cholera organisms was computed via the trapezoidal rule.
Time Frame: Day 1 to Day 5 (prior to first dose of antibiotic)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: liters * hours
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
liters * hours | 14.91 [9.3 to 20.8] | 13.80 [9.3 to 17.7]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.5992, Van Elteren test; Stratified by blood type group; Difference in Median = 1.1, 95% CI 2-sided [-4.5 to 7.8]

7. Secondary Outcome: Peak Shedding of Cholera Organisms
Description: Quantitative cultures were performed on the first two stool samples of each 24-hour period prior to the initiation of antibiotics to determine the number of cholera organisms per gram of stool. Peak shedding represents the highest colony-forming unit (CFU) counts observed for each participant.
Time Frame: Day 1 to Day 5 (prior to first dose of antibiotic)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CFU/g
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
CFU/g | 124960186.25 (163145761.682) | 186793500.00 (304578375.607)

8. Secondary Outcome: Duration of Diarrheal Episodes
Description: Duration of diarrheal episodes was calculated using Kaplan-Meier methods as the time from cholera challenge to the time of the first formed stool (Grade 1), after which all following stools were also formed.
Time Frame: Day 1 to Day 5 (prior to first dose of antibiotics)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
hours | 156.48 [114.1 to 217.8] | 169.68 [108.9 to 216.4]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.6527, Log Rank; Stratified by blood type group

9. Secondary Outcome: Total Number of Loose (Grade 3-5) Stools
Description: Total number of loose stools (Grade 3 and above) per participant during the interval immediately following challenge and prior to initiation of antibiotic therapy.
Time Frame: Day 1 to Day 5 (prior to first dose of antibiotic therapy)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: loose stools
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
loose stools | 12.0 [5 to 15] | 10.5 [8 to 18]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.5377, Van Elteren test; Stratified by blood type group; Difference in Median = 1.5, 95% CI 2-sided [-7.0 to 5.5]

10. Secondary Outcome: Percentage of Participants With Fever Following Cholera Challenge
Description: The presence of fever was defined as a body temperature of ≥ 39°C (102.1°F).
Time Frame: Day 1 to Day 5, prior to first dose of antibiotics
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
percentage of participants | 6.3 [0.2 to 30.2] | 5.0 [0.1 to 24.9]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.8705, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, stratified by blood type group; Difference = 1.3, 95% CI 2-sided [-14.0 to 16.5]

11. Secondary Outcome: Percentage of Participants With Vomiting Following Cholera Challenge
Time Frame: Day 1 to Day 5, prior to first dose of antibiotics
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 16 | 20
percentage of participants | 6.3 [0.2 to 30.2] | 25.0 [8.7 to 49.1]
Statistical Analysis 1: Comparison: iOWH032 vs Placebo; Test type: Superiority; p = 0.1404, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, stratified by blood type group; Difference = -18.8, 95% CI 2-sided [-41.1 to 3.6]

12. Secondary Outcome: Number of Participants With Solicited Adverse Effects
Description: Solicited adverse events (AEs) include nausea, abdominal discomfort and pain, abdominal cramps, headache, malaise, anorexia, pollakiuria, micturition urgency, sinus tachycardia, increased alertness, and were collected by interview through 7 days post-challenge (Days 1-8)
Time Frame: Day 1 - Day 8
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  Any solicited adverse event | 3 | 2
  Abdominal discomfort | 2 | 0
  Headache | 1 | 0
  Malaise | 0 | 1
  Nausea | 0 | 1

13. Secondary Outcome: Number of Participants With Unsolicited Treatment-emergent Adverse Events (TEAE)
Description: Unsolicited AEs include any AEs reported spontaneously by the participant, observed by the study personnel during study visits or those identified during review of medical records or source documents. Investigators assigned causality of unsolicited AEs to either the study drug, cholera infection, or an alternate etiology.
Time Frame: From first dose of study drug up to Day 29
Population: All participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | iOWH032 | Placebo
Number analyzed (Participants) | 23 | 24
Participants
  Any unsolicited TEAE | 18 | 21
  Study drug-related TEAE | 4 | 3
  TEAE leading to discontinuation from study | 0 | 0
  TEAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events and deaths were collected from first dose of study drug up to Day 180. Non-serious adverse events are reported from first dose of study drug up to Day 29.
Arm/Group | iOWH032 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/24
Other Adverse Events (participants affected / at risk) | 18/23 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | iOWH032 (N=23) | Placebo (N=24)
Pyelonephritis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | iOWH032 (N=23) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 1 | 6
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Haematochezia (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 5
Chills (General disorders) | 4 | 2
Pain (General disorders) | 1 | 3
Chest discomfort (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 9
Dizziness (Nervous system disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3
Blood potassium decreased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Full blood count increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 6 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Candida infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04150250/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04150250/SAP_001.pdf